CLINICAL TRIAL: NCT03056378
Title: Phase I Clinical Trial of Pooled Red Blood Cells for Transfusion
Brief Title: POOLED Red Blood Cells Prepared From Pooling 5 Leukoreduced, Irradiated RBC Units
Acronym: Pooled RBCs
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No patients enrolled. Study withdrawn.
Sponsor: New York Blood Center (Other)
Collaborators: Westchester Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NYBC-0088
Record Dates: First submitted 2017-01-13; First posted 2017-02-17 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Transfusion Reaction; Anemia
MeSH Terms: conditions — Transfusion Reaction; Anemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pooled RBCs (Experimental): Transfusion of an investigational transfusion blood component: POOLED-RBCs Phenotype matched/ compatible for ABO, D, C, E, and K (blood type of pool will be match patient's type), leukoreduced, and irradiated
  Interventions: Biological: Standard RBCs
- Standard RBCs (Active Comparator): Transfusion of standard transfusion blood component: additive solution leukoreduced, irradiated RBC product Phenotype matched/ compatible for ABO, D, C, E, and K (blood type of pool will be match patient's type)
  Interventions: Biological: Standard RBCs

INTERVENTIONS:
Biological: Standard RBCs — Transfusion of standard pRBCs that are matched for C, E and K

SUMMARY:
The purpose of the study is to determine the safety of pooled red blood cells (RBCs) compared to standard leukoreduced RBC products stored in additive solution. The primary objective is to determine if there is no significant difference in transfusion associated adverse events in POOLED-RBCs compared to standard RBC product groups. Secondarily to determine if there are no significant differences in new antibody and new positive direct antiglobulin test (DAT) formation in the POOLED-RBCs compared to standard RBC product groups.

DETAILED DESCRIPTION:
This research study is enrolling subjects who are receiving RBC (red blood cell) blood transfusions as part of their treatment. In this study, we are testing a new way of preparing RBC units (pooled RBC units) for transfusion compared to the standard RBC units. We are testing this because blood transfusions may be associated with side effects that may be harmful. We have developed a new way to process RBC for transfusion to try and reduce some of those side effects.

The pooled RBC units will be made by sterilely pooling five (5) single RBC units into one container where the blood will be mixed together, and then separated into five individual RBC units, ready to be used for transfusion. The purpose of the study is to determine the safety of the blood prepared in this new way compared to standard RBC products.

The primary objective is to determine if there is no significant difference in transfusion associated adverse events in POOLED-RBCs compared to standard RBC product groups. Secondarily to determine if there are no significant differences in new antibody and new positive direct antiglobulin test (DAT) formation in the POOLED-RBCs compared to standard RBC product groups.

ELIGIBILITY:
Inclusion Criteria:

* Age>= 18 years
* Hematology/ oncology or other chronic transfusion dependent patients
* Patients who are in need of transfusion due to low hemoglobin level (<8 gm/dl)
* Patients who only require one or two transfusion episode of 1-2 RBC units each during 60 day period
* Currently not planning to be pregnant during the study period

Exclusion Criteria:

* Previously identified alloantibodies (other than to D, C, E and K)
* Positive direct antiglobulin test, currently or within the last year
* Emergency transfusion
* Patients < 18 years old
* Need for specialized products, such as washed
* Patients involved in other RBC transfusion clinical trial
* Currently or planning to be pregnant within the proposed study period

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Quantitation of adverse events | 60 day endpoint

SECONDARY OUTCOMES:
Quantitation of RBC alloantibody formation | 15 and 30 minutes post-transfusion
  Quantitation of new DAT formation

CONTACTS AND LOCATIONS:
Overall Officials: Beth Shaz, M.D., Principal Investigator — New York Blood Center
Locations (1):
- Westchester Medical Center/New York Medical College, Valhalla, New York, United States

REFERENCES:
- [Background] Hendrickson JE, Hillyer CD. Noninfectious serious hazards of transfusion. Anesth Analg. 2009 Mar;108(3):759-69. doi: 10.1213/ane.0b013e3181930a6e. PMID 19224780
- [Background] Tobian AA, Fuller AK, Uglik K, Tisch DJ, Borge PD, Benjamin RJ, Ness PM, King KE. The impact of platelet additive solution apheresis platelets on allergic transfusion reactions and corrected count increment (CME). Transfusion. 2014 Jun;54(6):1523-9; quiz 1522. doi: 10.1111/trf.12498. Epub 2013 Nov 19. PMID 24251374
- [Background] Hess JR; Biomedical Excellence for Safer Transfusion (BEST) Collaborative. Scientific problems in the regulation of red blood cell products. Transfusion. 2012 Aug;52(8):1827-35. doi: 10.1111/j.1537-2995.2011.03511.x. Epub 2012 Jan 9. PMID 22229278
- [Background] Marthur A, Stassinopoulos A, Hess JR, Narla M, Shaz BH. Effects of pooling multiple red blood cell units to improve storage. Blood 2012;120:3437
- [Background] Mathur A, Chowdhury R, Hillyer CD, Mitchell WB, Shaz BH. Storage characteristics of multiple-donor pooled red blood cells compared to single-donor red blood cell units. Transfusion. 2016 Dec;56(12):2941-2947. doi: 10.1111/trf.13866. Epub 2016 Oct 5. PMID 27704557
- [Background] Lasalle-Williams M, Nuss R, Le T, Cole L, Hassell K, Murphy JR, Ambruso DR. Extended red blood cell antigen matching for transfusions in sickle cell disease: a review of a 14-year experience from a single center (CME). Transfusion. 2011 Aug;51(8):1732-9. doi: 10.1111/j.1537-2995.2010.03045.x. Epub 2011 Feb 18. PMID 21332724
- [Background] Verduin EP, Brand A, Schonewille H. Is female sex a risk factor for red blood cell alloimmunization after transfusion? A systematic review. Transfus Med Rev. 2012 Oct;26(4):342-53, 353.e1-5. doi: 10.1016/j.tmrv.2011.12.001. Epub 2012 Jan 13. PMID 22244869
- [Background] Custer B, Agapova M, Martinez RH. The cost-effectiveness of pathogen reduction technology as assessed using a multiple risk reduction model. Transfusion. 2010 Nov;50(11):2461-73. doi: 10.1111/j.1537-2995.2010.02704.x. PMID 20497512
- [Background] Sweeney JD, Kouttab NM, Holme S, Kurtis JD, Cheves TA, Nelson EJ. Prestorage pooled whole-blood-derived leukoreduced platelets stored for seven days, preserve acceptable quality and do not show evidence of a mixed lymphocyte reaction. Transfusion. 2004 Aug;44(8):1212-9. doi: 10.1111/j.1537-2995.2004.03438.x. PMID 15265126
- [Background] Thiele T, Heddle N, Greinacher A. Donor exposures in recipients of pooled platelet concentrates. N Engl J Med. 2013 Jan 31;368(5):487-9. doi: 10.1056/NEJMc1213383. No abstract available. PMID 23363522
- [Background] Zou S, Stramer SL, Dodd RY. Donor testing and risk: current prevalence, incidence, and residual risk of transfusion-transmissible agents in US allogeneic donations. Transfus Med Rev. 2012 Apr;26(2):119-28. doi: 10.1016/j.tmrv.2011.07.007. Epub 2011 Aug 25. PMID 21871776
- [Background] Stramer SL, Notari EP, Krysztof DE, Dodd RY. Hepatitis B virus testing by minipool nucleic acid testing: does it improve blood safety? Transfusion. 2013 Oct;53(10 Pt 2):2449-58. doi: 10.1111/trf.12213. Epub 2013 Apr 23. PMID 23607261
- [Background] Levin AE, Williamson PC, Bloch EM, Clifford J, Cyrus S, Shaz BH, Kessler D, Gorlin J, Erwin JL, Krueger NX, Williams GV, Penezina O, Telford SR 4th, Branda JA, Krause PJ, Wormser GP, Schotthoefer AM, Fritsche TR, Busch MP. Serologic screening of United States blood donors for Babesia microti using an investigational enzyme immunoassay. Transfusion. 2016 Jul;56(7):1866-74. doi: 10.1111/trf.13618. Epub 2016 May 25. PMID 27224258
- [Background] Levin AE, Williamson PC, Erwin JL, Cyrus S, Bloch EM, Shaz BH, Kessler D, Telford SR 3rd, Krause PJ, Wormser GP, Ni X, Wang H, Krueger NX, Caglioti S, Busch MP. Determination of Babesia microti seroprevalence in blood donor populations using an investigational enzyme immunoassay. Transfusion. 2014 Sep;54(9):2237-44. doi: 10.1111/trf.12763. Epub 2014 Jul 4. PMID 24995863
- [Background] Tormey CA, Sweeney JD, Champion MH, Pisciotto PT, Snyder EL, Wu Y. Analysis of transfusion reactions associated with prestorage-pooled platelet components. Transfusion. 2009 Jun;49(6):1242-7. doi: 10.1111/j.1537-2995.2009.02128.x. Epub 2009 Mar 23. PMID 19389029
- [Background] Daurat A, Roger C, Gris J, Daurat G, Feissel M, Le Manach Y, Lefrant J, Muller L. Apheresis platelets are more frequently associated with adverse reactions than pooled platelets both in recipients and in donors: a study from French hemovigilance data. Transfusion. 2016 Jun;56(6):1295-303. doi: 10.1111/trf.13475. Epub 2016 Jan 26. PMID 26814984
- See also: National Healthcare Safety Network Biovigilance component Hemovigilance module Surveillance Protocol: Center for Disease Control Prevention, ed.2017 — https://www.cdc.gov/nhsn/pdfs/biovigilance/bv-hv-protocol-current.pdf